CLINICAL TRIAL: NCT03919045
Title: Saline Injections for Prophylactic Treatment of Chronic Migraine - a Randomized Controlled Study
Brief Title: Saline Injections for Prophylactic Treatment of Chronic Migraine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to Covid-19 the rehabilitation unit where the trial was conducted were closed and the trial active clinician had to work at the hospital intensive care.
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Migraine1; 2018-003868-32 (EudraCT Number)
Record Dates: First submitted 2019-04-08; First posted 2019-04-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Migraine
Keywords: Chronic migraine; Saline injection
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: No Outcome assessor present in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium chloride injection (Experimental): Sodium chloride 9mg/ml by injection
  Interventions: Drug: Saline injection
- Needle sting (Placebo Comparator): Brief needle stings without injection
  Interventions: Procedure: Placebo

INTERVENTIONS:
Drug: Saline injection — Half of the patients will be randomized to saline injections into the neck and head muscles
  Other Names: Sodium chloride Braun; Sodium chloride Fresenius Krabi
  Arms: Sodium chloride injection
Procedure: Placebo — Half of the group will be treated with needle stings without injections
  Arms: Needle sting

SUMMARY:
In this study, the investigators want to investigate whether saline injections in the neck and head muscles can reduce symptoms of chronic migraine. In existing studies, saline injections (used as placebo treatment) have given patients with chronic migraine an average of 7 headache-free days per month.

DETAILED DESCRIPTION:
Patients who meet the diagnostic criteria for chronic migraine will be invited to participate in the study. All participants will undergo a medical examination. The participants will fill out an electronic headache diary for one month. This will give a picture of the current headache pattern and establish a baseline. The participants will then be randomized into two groups: saline injections or needle sticks without injection. They will not be aware of which group they belong to. The treatment will be repeated on two occasions three months apart. The headache diary will continue during the treatment period and up to three months after the second treatment. The effect will be analyzed by comparing baseline data from the headache diary to data after treatment. The primary outcome of the study is the number of days with headache, during a 28-day period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the diagnostic criteria for chronic migraine (headache that have occurred on at least 15 days per month, for at least three months. At least eight of the headache episodes must be typical for migraine).
* Participants must be able to understand and give informed consent to participate in the study.
* Participants must be aged 18-65 years.

Exclusion Criteria:

* Participants must not suffer from other medical conditions that may affect the outcome of the study, including Horton's headache, temporal arteritis, trigeminal neuralgia, chronic paroxysmal hemi-crania, atypical facial pain and headache of unknown cause.
* Participants must not have medical conditions that require use of drugs that can affect the headache pattern (for example rheumatic disorders).
* Participants must not suffer from malignant diseases.
* Participants must not plan to make changes to existing prophylactic headache medication during the study. Patients may, if already on treatment, choose to continue this throughout the course of the study, or choose to stop the prophylactic treatment at least one week before the start of the baseline period.
* Participants must not have an ongoing patient-doctor contact with the physician giving the injections.
* Participants must not have an ongoing patient-doctor contact with the monitor of the study.
* Participants must not have received injection therapy in the face, head or neck muscles (medical or cosmetic) less than three months before the start of the study, nor should they plan such treatment during the course of the study.
* Participants must not be pregnant or plan pregnancy during the course of the study.
* Participants must not breastfeed or plan to do so during the study.
* Participants must not have any contraindications to injection therapy (such as disease with increased bleeding tendency or treatment with certain types of blood thinners).
* Participants must have no difficulty understanding or making themselves understood in Swedish.
* Participants must be able to fill out the headache diary and questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Change in number of Days with headache | change between baseline 28 day period prior injection1 and 28 day period ending study
  A headache day is defined as: 1) a day with headache ≥ 4 hours or 2) a day with headache of any duration, where the headache is relieved with acute headache medication (AHM)
  By AHM is meant a drug that is taken when needed for the purpose of relieving headaches, including any of the following:
  * Paracetamol
  * Aspirin
  * NSAID
  * Triptan
  * Opioid
  * Ergotamine
  * Dihydroergotamine
  The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.
Change in number of Days with headache | change between baseline and the 28-day period preceding the second injection
  A headache day is defined as: 1) a day with headache ≥ 4 hours or 2) a day with headache of any duration, where the headache is relieved with acute headache medication.
  By AHM is meant a drug that is taken when needed for the purpose of relieving headaches, including any of the following:
  * Paracetamol
  * Aspirin
  * NSAID
  * Triptan
  * Opioid
  * Ergotamine
  * Dihydroergotamine
  The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.

SECONDARY OUTCOMES:
Number of Days with moderate or severe headache | change between baseline 28 day period prior injection1 and 28 day period ending study
  A headache day with moderate or severe intensity is defined as: 1) a day with headache ≥ 4 hours and with a peak of moderate or severe intensity or 2) a day with headache of any duration or intensity, where the headache is relieved with AHM. The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.
Number of Days with moderate or severe headache | change between baseline and the 28-day period preceding the second injection
  A headache day with moderate or severe intensity is defined as: 1) a day with headache ≥ 4 hours and with a peak of moderate or severe intensity or 2) a day with headache of any duration or intensity, where the headache is relieved with AHM. The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.
Number of days with acute headache medication | change between baseline 28 day period prior injection1 and 28 day period ending study
  Number of days the respondent stated that AHM has been taken.The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.
Number of days with acute headache medication | change between baseline and the 28-day period preceding the second injection
  Number of days the respondent stated that AHM has been taken.The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.
Number of days with acute headache medication that requires prescription | change between baseline 28 day period prior injection1 and 28 day period ending study
  Number of days the respondent stated that he or she has taken acute headache medication that require prescription, ie all drugs in the list in primary outcome above that require prescription by a doctor.The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.
Number of days with acute headache medication that requires prescription | change between baseline and the 28-day period preceding the second injection
  Number of days the respondent stated that he or she has taken acute headache medication that require prescription, ie all drugs in the list in primary outcome above that require prescription by a doctor.The primary efficacy measure is the change between the baseline 28-day period (4 weeks prior injection 1) and the corresponding period during follow-up, i.e. the 28-day period ending the study. a secondary efficacy measure is the change between the baseline and the 28-day period preceding the second injection.
Change in outcome of disease-specific quality of Life: Migraine-specific Quality of Life Questionnaire (MSQ v2.1) | Change between baseline and 12 weeks after second injection
  Change in Migraine-specific Quality of Life Questionnaire (MSQ v2.1)
Change in outcome of disease-specific implications: Headache Impact Test (HIT-6) | Change between baseline and 12 weeks after second injection
  Change in Headache Impact Test (HIT-6)

CONTACTS AND LOCATIONS:
Overall Officials: Malin Kim, MD, Principal Investigator — Rehabilitation clinic, Southern Älvsborg Hospital
Locations (1):
- Rehabilitation clinic, Southern Älvsborg Hospital, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole JC, Lin P, Rupnow MF. Validation of the Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQ v. 2.1) for patients undergoing prophylactic migraine treatment. Qual Life Res. 2007 Sep;16(7):1231-7. doi: 10.1007/s11136-007-9217-1. Epub 2007 Apr 28. PMID 17468941
- [Background] Dodick DW, Turkel CC, DeGryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: pooled results from the double-blind, randomized, placebo-controlled phases of the PREEMPT clinical program. Headache. 2010 Jun;50(6):921-36. doi: 10.1111/j.1526-4610.2010.01678.x. Epub 2010 May 7. PMID 20487038
- [Background] Freitag FG, Diamond S, Diamond M, Urban G. Botulinum Toxin Type A in the treatment of chronic migraine without medication overuse. Headache. 2008 Feb;48(2):201-9. doi: 10.1111/j.1526-4610.2007.00963.x. Epub 2007 Nov 28. PMID 18042229
- [Background] Gandek B, Alacoque J, Uzun V, Andrew-Hobbs M, Davis K. Translating the Short-Form Headache Impact Test (HIT-6) in 27 countries: methodological and conceptual issues. Qual Life Res. 2003 Dec;12(8):975-9. doi: 10.1023/a:1026171315263. PMID 14651416
- [Background] Smelt AF, Assendelft WJ, Terwee CB, Ferrari MD, Blom JW. What is a clinically relevant change on the HIT-6 questionnaire? An estimation in a primary-care population of migraine patients. Cephalalgia. 2014 Jan;34(1):29-36. doi: 10.1177/0333102413497599. Epub 2013 Jul 10. PMID 23843470
- [Background] Goadsby PJ. Migraine pathophysiology. Headache. 2005 Apr;45 Suppl 1:S14-24. doi: 10.1111/j.1526-4610.2005.4501003.x. PMID 15833086
- [Background] Kim M, Danielsson A, Ekelund A-C, Kemppainen E, Sjögren P, Svanberg T, Szalo G,Samuelsson O. Title:Botulinum toxin type A for Prophylactic Treatment of Chronic Migraine [Botulinum toxin typ Asom profylaktisk behandling av kronisk migrän]. Göteborg: Västra Götalandsregionen, SahlgrenskaUniversitetssjukhuset, HTA-centrum; 2014. Regional activity-based HTA 2014:70